CLINICAL TRIAL: NCT07343531
Title: A Prospective Phase II Study Of Moderately Hypo-Fractionated External-beam Radiotherapy With Concurrent Chemotherapy and High Dose Rate Brachytherapy In Cervical Cancer
Brief Title: A Study Of Moderately Hypo-Fractionated External-beam Radiotherapy With Concurrent Chemotherapy and High Dose Rate Brachytherapy In Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD221/2025
Record Dates: First submitted 2026-01-01; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Cervical Carcinoma Stage III; Cervical Carcinoma Stage IIB; Cervical Carcinoma Stage II
Keywords: cervical cancer hypofractionation EBRTH
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective single-arm clinical trial to assess the clinical response, acute and a two-year late toxicities of moderately hypo-fractionated external-beam radiotherapy with concurrent chemotherapy and high-dose rate brachytherapy in cervical cancer.
  A phase II trial for patients histopathologically diagnosed as invasive cervical carcinoma with above mentioned eligibility criteria recruited from the gynecological oncology outpatient unit of a single center in Egypt, at the clinical oncology and nuclear medicine department, Ain Shams University Hospital.
  The trial is a single-arm study (experimental group ): 30 patients will receive external beam radiotherapy (EBRT) 40 Gy / 16 fractions with additional 6:10 Gy boost on positive pelvic L.Ns if found either sequential or simultaneous integrated boost (SIB) (according to patient tolerability) with IMRT or VMAT technique followed by High-dose rate (HDR) Brachytherapy 28 Gy /4 fractions 7 Gy per fraction over 2 weeks .
Masking Description: The primary endpoint:
  - The tumor response rate on Magnetic resonance imaging (MRI) images will be graded as proposed in Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) to be done before start of the radiotherapy, at the last week of external beam radiotherapy and at 3 month-follow up visits then at regular follow up.
  The secondary endpoints :
  1-Acute and a two-year late toxicities are assessed by clinical assessment during each follow-up appointment, and scored according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 . Clinically relevant toxicities of gastrointestinal, genitourinary, vaginal and non-specific general symptoms (i.e. fatigue, malaise and pain) will be collected. Haematological disorders will also be collected through weekly blood work checks. Acute toxicities will be collected at baseline, and then weekly during radiotherapy/chemoradiotherapy and at 3 months after completion of radiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): 30 patients will receive external beam radiotherapy (EBRT) 40 Gy / 16 fractions with additional 6:10 Gy boost on positive pelvic L.Ns if found either sequential or simultaneous integrated boost (SIB) (according to patient tolerability) with IMRT or VMAT technique followed by High-dose rate (HDR) Brachytherapy 28 Gy /4 fractions 7 Gy per fraction over 2 weeks
  Interventions: Radiation: moderate hypofractionation external beam radiotherapy

INTERVENTIONS:
Radiation: moderate hypofractionation external beam radiotherapy — 30 patients will receive external beam radiotherapy (EBRT) 40 Gy / 16 fractions with additional 6:10 Gy boost on positive pelvic L.Ns if found either sequential or simultaneous integrated boost (SIB) (according to patient tolerability) with IMRT or VMAT technique followed by High-dose rate (HDR) Brachytherapy 28 Gy /4 fractions 7 Gy per fraction over 2 weeks.Concurrent weekly cisplatin 40 mg/m2 will be received .
  -Concurrent weekly carboplatin AUC 2 will be received if cisplatin is not tolerated (creatinine clearance 40:60 ml/min) .
  HDR brachytherapy boost will be given 28 Gy/ 4 fractions 7 Gy per fraction over 2 weeks to be started within a week after the end of external beam radiotherapy sessions.

SUMMARY:
Cancer of the uterine cervix is one of the most common gynecologic cancer diagnosis and cause of death among gynecologic cancers worldwide .The two major histologic types of cervical cancer are squamous cell carcinoma, adenocarcinoma and the preinvasive disease that corresponds with these histologies share many of the same risk factors .

Cancer cervix can be treated definitively with concurrent chemoradiation (external beam radiotherapy and chemotherapy) followed by high dose rate brachytherapy. Treatment duration can be shortened by increasing the dose per fraction of treatment, which can improve survival rates, reduce the risk of treatment failure, reduce costs and patient exposure.

DETAILED DESCRIPTION:
The objective of this study is: to assess the clinical response (as a primary endpoint), acute and a two-year late toxicities (as a secondary endpoint) of moderately hypo-Fractionated external-beam radiotherapy with concurrent chemotherapy and high-dose rate brachytherapy in cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. International Federation of Gynecology and Obstetrics (FIGO) IB1 cervical cancers if not surgical candidates, but amenable to definitive chemoradiotherapy.
3. FIGO Stage IB2, IB3, IIA or IIB cervical cancers
4. FIGO stage IIIA, IIIB.
5. FIGO stage IIIC1 cervical cancers are candidates but must meet all the following criteria (to avoid extented field technique ): The largest radiologically suspicious positive pelvic node is less than 3 cm. Less than 3 radiologically suspicious positive nodes. No suspicious nodes located in the common iliac chain.
6. Histologically-confirmed invasive uterine cervical carcinoma of subtypes squamous cell, adenocarcinoma or adenosquamous cell.
7. Candidate for definitive chemoradiotherapy to be delivered with weekly cisplatin (Creatinine clearance more than 60 ml/min). Carboplatin AUC 2 is acceptable alternative if cisplatin is not tolerated (creatinine clearance 40:60 ml/min) .
8. Brachytherapy candidate.
9. Eastern Cooperative Oncology Group (ECOG) performance status up to 2 .

Exclusion Criteria:

* 1.FIGO stage IA, IIIC2, IVA or IVB. 2.FIGO stage IIIC1 with node is equal or greater than 3 cm, common iliac node or greater than 2 radiologically suspicious nodes.

  3.Previous pelvic or abdominal radiotherapy. 4.Active inflammatory bowel disease. 5.Active connective tissue disorder (eg. scleroderma, systemic lupus erythematous).

  6.Patient unable to undergo MR scan 7.Eastern Cooperative Oncology Group (ECOG) performance status equal to 3 or more.

  8.Creatinine clearance less than 40 ml/min.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
tumor response rate | two years
  The tumor response rate on Magnetic resonance imaging (MRI) images will be graded as proposed in Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) to be done before start of the radiotherapy, at the last week of external beam radiotherapy and at 3 month-follow up visit then at regular follow up visits

SECONDARY OUTCOMES:
acute toxicity | 3 months
  Acute toxicities are assessed by clinical assessment during each follow-up appointment, and scored according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 . Clinically relevant toxicities of gastrointestinal, genitourinary, vaginal and non-specific general symptoms (i.e. fatigue, malaise and pain) will be collected. Haematological disorders will also be collected through weekly blood work checks. Acute toxicities will be collected at baseline, and then weekly during radiotherapy/chemoradiotherapy and at 3 months after completion of radiotherapy
Late toxicity | 2 years
  Late toxicities are assessed by clinical assessment during each follow-up appointment, and scored according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 . Clinically relevant toxicities of gastrointestinal, genitourinary, vaginal and non-specific general symptoms (i.e. fatigue, malaise and pain) will be collected. Late toxicities will be collected at 3 months after completion of radiotherapy till 2 years
Progression free survival | 2 years
  Progression-free survival is defined as time from the date of treatment initiation to the date of progression, date of death from any cause, or date of last follow-up, whichever occurs first. Cancer progression can be identified during physical examination ,EUA ,clinically by imaging of any kind or biopsy within a time frame of 2 years .
Overall survival | 2 years
  Overall survival is defined as time from date of treatment initiation to death from any reason or last follow-up ,whichever occurs first, with a time frame of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University, Cairo, Cairo Governorate, Egypt